CLINICAL TRIAL: NCT00711009
Title: A Randomized, Open-label Study of Lopinavir/Ritonavir 400/100 mg Tablet Twice Daily + Co-formulated Emtricitabine/Tenofovir Disoproxil Fumarate 200/300 mg Once Daily Versus Lopinavir/Ritonavir 400/100 mg Tablet Twice Daily + Raltegravir 400 mg Twice Daily in Antiretroviral Naive, HIV-1 Infected Subjects
Brief Title: Study Comparing Lopinavir/Ritonavir (LPV/r) + Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) With a Nucleoside Sparing Regimen Consisting of Lopinavir/Ritonavir + Raltegravir (RAL)
Acronym: PROGRESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M10-336; 2008-000881-22 (EudraCT Number)
Record Dates: First submitted 2008-07-03; First posted 2008-07-08 (Estimated); Results first posted 2011-02-02 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Human Immunodeficiency Virus Infection
Keywords: Human Immunodeficiency Virus infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Lopinavir; lopinavir-ritonavir drug combination; Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Raltegravir Potassium

ARMS (2):
- LPV/r + FTC/TDF (Active Comparator): lopinavir/ritonavir 400/100 milligram (mg) tablet twice-daily + co-formulated emtricitabine/tenofovir disoproxil fumarate 200/300 mg once-daily
  Interventions: Drug: lopinavir/ritonavir (LPV/r); Drug: emtricitabine/tenofovir disoproxil fumarate (FTC/TDF)
- LPV/r + RAL (Experimental): lopinavir/ritonavir 400/100 mg tablet twice-daily + raltegravir 400 mg twice-daily
  Interventions: Drug: lopinavir/ritonavir (LPV/r); Drug: raltegravir (RAL)

INTERVENTIONS:
Drug: lopinavir/ritonavir (LPV/r) — LPV/r 400/100 mg BID
  Other Names: ABT-378; lopinavir/ritonavir; LPV/r; Kaletra
Drug: emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) — FTC/TDF 200/300 mg QD
  Other Names: emtricitabine/tenofovir disoproxil fumarate; FTC/TDF; Truvada
  Arms: LPV/r + FTC/TDF
Drug: raltegravir (RAL) — RAL 400 mg BID
  Other Names: raltegravir; RAL; Isentress; MK-0518
  Arms: LPV/r + RAL

SUMMARY:
The purpose of this study is to compare the safety, tolerability, and antiviral activity of the lopinavir/ritonavir tablet when administered in combination with reverse transcriptase inhibitors to lopinavir/ritonavir tablets when administered in combination with a human immunodeficiency virus type 1 ( HIV-1) integrase inhibitor in antiretroviral naive HIV-1 infected subjects.

ELIGIBILITY:
Inclusion Criteria:

* Participants must provide written, voluntary informed consent to participate in the study.
* Participants must be naive to antiretroviral treatment with HIV RNA greater than or equal to 1,000 copies/mL at screening, and in the investigator's opinion, require antiretroviral therapy.
* Participant's vital signs, physical examination, and laboratory results must not exhibit evidence of acute illness.
* Participant has not been treated for an active acquired immune deficiency syndrome (AIDS)-defining opportunistic infection within 45 days of initiating study drug. Participants who are on stable maintenance therapy for an opportunistic infection may be enrolled after consultation with the Sponsor.
* Participant does not require and agrees not to take any drugs that are contraindicated or have significant pharmacokinetic interactions with study drugs during the course of the study. Participant agrees not to take any medication during the study, including over-the-counter medicines, vitamins, minerals, herbal preparations, alcohol, or recreational drugs without the knowledge and permission of the principal investigator.
* Female participants must be either postmenopausal for at least one year, surgically sterile, or must use a non-hormonal method of birth control that is acceptable to both the participant and investigator. All female participants must have a urine pregnancy test performed at screening visit and on Day minus 1/baseline, and results of both tests must be negative. Female participants may not be breastfeeding.
* Participants have received no prior treatment with an HIV-1 integrase inhibitor.

Exclusion Criteria:

* Participants must not have history of an allergic reaction or significant sensitivity to the study drugs.
* Participants may not have an ongoing history of substance abuse or psychiatric illness that could preclude protocol adherence.
* Participant cannot have resistance to lopinavir/ritonavir, tenofovir, or emtricitabine based on the HIV-1 drug resistance genotypic test results at the screening visit.
* Participant may not have significant medical history of concomitant illness or disease that would adversely affect his/her participating in the study.
* Participants may not have received any investigational drug or investigational vaccine within 30 days prior to study drug administration.
* Participants may not have any of the following abnormal screening results: Hemoglobin <= 8.0 grams/deciliter, absolute neutrophil count <= 750 cells/microliter, Platelet count <= 50,000 per milliliter, alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) or aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) >= 3.0 x upper limit of normal (ULN), calculated creatinine clearance < 50 milliliter/minute, hepatitis B surface antigen (HBsAg) is positive.
* The investigator considers the participant to be an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2008-07; Primary Completion 2009-11 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Podsadecki, MD, Study Director — Abbott
Locations (37):
- United States (14):
  - Site Reference ID/Investigator# 8431, Phoenix, Arizona
  - Site Reference ID/Investigator# 8432, Beverly Hills, California
  - Site Reference ID/Investigator# 8394, Atlantis, Florida
  - Site Reference ID/Investigator# 8393, Ft. Pierce, Florida
  - Site Reference ID/Investigator# 8425, Orlando, Florida
  - Site Reference ID/Investigator# 8402, Tampa, Florida
  - Site Reference ID/Investigator# 8396, Vero Beach, Florida
  - Site Reference ID/Investigator# 8395, Atlanta, Georgia
  - Site Reference ID/Investigator# 8429, Decatur, Georgia
  - Site Reference ID/Investigator# 8424, Boston, Massachusetts
  - Site Reference ID/Investigator# 8426, Charlotte, North Carolina
  - Site Reference ID/Investigator# 11461, Huntersville, North Carolina
  - Site Reference ID/Investigator# 8403, Dallas, Texas
  - Site Reference ID/Investigator# 8433, Houston, Texas
- Canada (4):
  - Site Reference ID/Investigator# 7963, Ottawa, Ontario
  - Site Reference ID/Investigator# 7831, Toronto, Ontario
  - Site Reference ID/Investigator# 7959, Toronto, Ontario
  - Site Reference ID/Investigator# 8099, Montreal, Quebec
- France (4):
  - Site Reference ID/Investigator# 7695, Lyon
  - Site Reference ID/Investigator# 7960, Montpellier
  - Site Reference ID/Investigator# 8063, Paris
  - Site Reference ID/Investigator# 7821, Paris
- Italy (4):
  - Site Reference ID/Investigator# 8052, Genoa
  - Site Reference ID/Investigator# 7789, Milan
  - Site Reference ID/Investigator# 8051, Perugia
  - Site Reference ID/Investigator# 8050, Rome
- Site Reference ID/Investigator# 8221, Wroclaw, Poland
- Puerto Rico (2):
  - Site Reference ID/Investigator# 7713, Bayamón
  - Site Reference ID/Investigator# 7700, Ponce
- Spain (8):
  - Site Reference ID/Investigator# 11102, Barcelona
  - Site Reference ID/Investigator# 7697, Barcelona
  - Site Reference ID/Investigator# 7689, Barcelona
  - Site Reference ID/Investigator# 7692, L'Hospitalet de Llobregat
  - Site Reference ID/Investigator# 7698, Madrid
  - Site Reference ID/Investigator# 7693, Madrid
  - Site Reference ID/Investigator# 7691, Madrid
  - Site Reference ID/Investigator# 7690, Seville

REFERENCES:
- [Derived] Reynes J, Trinh R, Pulido F, Soto-Malave R, Gathe J, Qaqish R, Tian M, Fredrick L, Podsadecki T, Norton M, Nilius A. Lopinavir/ritonavir combined with raltegravir or tenofovir/emtricitabine in antiretroviral-naive subjects: 96-week results of the PROGRESS study. AIDS Res Hum Retroviruses. 2013 Feb;29(2):256-65. doi: 10.1089/aid.2011.0275. Epub 2012 Aug 3. PMID 22730929
- [Derived] Reynes J, Lawal A, Pulido F, Soto-Malave R, Gathe J, Tian M, Fredrick LM, Podsadecki TJ, Nilius AM. Examination of noninferiority, safety, and tolerability of lopinavir/ritonavir and raltegravir compared with lopinavir/ritonavir and tenofovir/ emtricitabine in antiretroviral-naive subjects: the progress study, 48-week results. HIV Clin Trials. 2011 Sep-Oct;12(5):255-67. doi: 10.1310/hct1205-255. PMID 22180523
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/search.cfm?startswith=Kaletra

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 additional participants were randomized but did not receive study drug and therefore were not included in the analyses.
Groups:
- LPV/r + FTC/TDF: lopinavir/ritonavir 400/100 mg tablet twice-daily + co-formulated emtricitabine/tenofovir disoproxil fumarate 200/300 mg once-daily
Period: Overall Study
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Started | 105 | 101
Completed | 90 | 82
Not Completed | 15 | 19
Not completed — Adverse Event/HIV-Related Event | 4 | 5
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 3 | 9
Not completed — Participant Noncompliant | 0 | 1
Not completed — Virologic Failure | 2 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Site closing | 0 | 1
Not completed — Dose adjustment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL | Total
Number analyzed (Participants) | 105 | 101 | 206
Age Continuous [Mean (Standard Deviation); unit: years] | 39.4 (11.24) | 39.8 (9.94) | 39.6 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 32
  Male | 86 | 88 | 174
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 22 | 44
  White | 81 | 74 | 155
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  North America | 61 | 59 | 120
  Europe | 44 | 42 | 86
Plasma Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) Level [Mean (Standard Deviation); unit: log10 copies/milliliter] | 4.3 (0.76) | 4.2 (0.83) | 4.2 (0.79)
CD4+ T-Cell Counts [Mean (Standard Deviation); unit: cells/microliter] | 297.6 (166.66) | 289.3 (149.03) | 293.5 (157.93)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Responding (Plasma HIV-1 Ribonucleic Acid [RNA] Levels Less Than 40 Copies/Milliliter [mL]) at Week 48 Based on the Food and Drug Administration (FDA) Time to Loss of Virologic Response (TLOVR) Algorithm
Description: A participant was classified as a responder at the first of 2 consecutive visits with plasma HIV-1 RNA levels below 40 copies/mL. The participant continued to be a responder until one of the following: the participant had 2 consecutive values greater than or equal to 40 copies/mL; the final measurement, if the final measurement was the first one documenting an increase in plasma HIV-1 RNA level to greater than or equal to 40 copies/mL; the participant discontinued participation in the study or died.
Time Frame: Baseline to Week 48
Population: Intent to treat (ITT) population, defined as all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 105 | 101
Percentage of Participants | 84.8 | 83.2
Statistical Analysis 1: Comparison: LPV/r + FTC/TDF vs LPV/r + RAL; The null hypothesis was that the response rate for the LPV/r + RAL arm was more than 20% lower than the response rate for the LPV/r + FTC/TDF arm. The planned sample size of 100 participants per treatment group provided 90% power to conclude that the LPV/r + RAL arm was non-inferior to the control arm, based on a non-inferiority margin of -20% (with a type I error rate of 0.05); Test type: Non-Inferiority or Equivalence — The exact 95% confidence interval for the difference in response rates (LPV/r + RAL minus LPV/r + FTC/TDF) was used to assess non-inferiority. The LPV/r+RAL arm was considered non-inferior to the LPV/r+FTC/TDF arm because the lower limit of the confidence interval was >/= -20%. Because the LPV/r+RAL arm was considered non-inferior based on the 20% margin, the results were assessed on a more rigorous 12% margin (-12%), as prespecified; p = 0.850, exact binomial method; Diff. in Percentage of Subj. Responding = -1.6, 95% CI 2-sided [-12.0 to 8.8]

2. Primary Outcome: Percentage of Participants With Moderate or Severe Treatment-emergent, Drug-related Adverse Events
Description: Treatment-emergent adverse events were defined as those occurring after study drug initiation and within 30 days after the last dose of study drug. Treatment-emergent, moderate or severe drug-related adverse events that occurred in at least 2% of participants in either treatment arm are presented.
Time Frame: Week 96
Population: Intent to treat (ITT) population, defined as all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 105 | 101
Percentage of participants
  Any adverse event | 34.3 | 30.7
  Diarrhoea | 16.2 | 7.9
  Hyperchloresterolaemia | 4.8 | 8.9
  Hypertriglyceridaemia | 2.9 | 5.9
  Hyperlipidaemia | 1.0 | 3.0
  Blood triglycerides increased | 1.9 | 3.0
  Alanine aminotransferase increased | 1.0 | 3.0
  Aspartate aminotransferase increased | 0 | 2.0
  Asthenia | 2.9 | 0

3. Secondary Outcome: Percentage of Participants Responding (Plasma HIV-1 RNA Levels Below 40 Copies/Milliliter [mL]) at Each Visit Based on the FDA Time to Loss of Virologic Response (TLOVR) Algorithm
Description: A participant was classified as a responder at the first of 2 consecutive visits with plasma HIV-1 RNA levels below 40 copies/mL. The participant continued to be a responder until one of the following: 1) the participant had 2 consecutive values greater than or equal to 40 copies/mL; the final measurement, if the final measurement was the first one documenting an increase in plasma HIV-1 RNA level to greater than or equal to 40 copies/mL; the participant discontinued participation in the study or died.
Time Frame: Baseline to Week 96
Population: Intention to treat analysis of all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 105 | 101
Percentage of Participants
  Week 2 | 7.6 | 33.7
  Week 4 | 17.1 | 63.4
  Week 8 | 36.2 | 75.2
  Week 16 | 67.6 | 81.2
  Week 24 | 80.0 | 83.2
  Week 32 | 85.7 | 85.1
  Week 40 | 84.8 | 87.1
  Week 48 | 84.8 | 83.2
  Week 60 | 82.9 | 75.2
  Week 72 | 78.1 | 71.3
  Week 84 | 74.3 | 70.3
  Week 96 | 68.6 | 66.3

4. Primary Outcome: Primary Outcome: Percentage of Participants With Potentially Clinically Significant Laboratory Values
Description: Potentially clinically significant laboratory values that occurred in at least 2% of participants in either treatment arm are presented.
Time Frame: Baseline to Week 96
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline laboratory value.
Measure: Number; unit: Percentage of participants
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 104 | 101
Percentage of participants
  Alananine aminotransferase >5x upper limit normal | 2.9 | 5.0
  Aspartate aminotransferase >5x upper limit normal | 2.9 | 5.0
  Creatinine phosphokinase >4x upper limit of normal | 8.7 | 19.8
  Calcium <1.75 millimoles/liter | 0 | 2.0
  Cholesterol >7.77 millimoles/liter | 13.5 | 16.8
  Triglycerides >8.475 millimoles/liter | 4.8 | 9.9
  Calc. creatinine clearance <50 milliliters/minute | 3.8 | 1.0
  Lipase >2x upper limit of normal | 7.7 | 4.0
  Neutrophils < 0.75 x 10^9/liter | 3.8 | 0
  Magnesium < 0.5 millimoles/liter | 0 | 2.0

5. Secondary Outcome: Mean Change in CD4+ T-Cell Counts From Baseline to Each Visit
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and the visit were included in the analysis of data at that visit. Number of participants in each visit analysis ranged from 98 and 96 participants in the LPV/r+FTC/TDF and LPV/r+RAL groups, respectively, at Week 8, to 80 and 76 participants in the LPV/r+FTC/TDF and LPV/r+RAL groups, respectively, at Week 96.
Measure: Mean (Standard Error); unit: cells/microliter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 105 | 101
cells/microliter
  Week 4 | 97.2 (10.94) | 113.4 (10.83)
  Week 8 | 107.9 (12.07) | 124.5 (12.20)
  Week 16 | 158.7 (13.94) | 141.6 (14.01)
  Week 24 | 154.9 (13.76) | 174.5 (13.99)
  Week 32 | 180.0 (13.42) | 188.2 (13.49)
  Week 40 | 204.6 (15.22) | 223.0 (15.55)
  Week 48 | 245.0 (18.02) | 241.9 (17.83)
  Week 60 | 243.4 (18.05) | 250.6 (18.45)
  Week 72 | 277.4 (20.10) | 269.9 (20.47)
  Week 84 | 309.6 (19.83) | 280.2 (21.05)
  Week 96 | 296.4 (20.38) | 281.0 (20.91)

6. Secondary Outcome: Time to Loss of Virologic Response - Percentage of Participants Still Categorized as Responders at Day 672
Description: Time of loss of virologic response was defined as the first of the following: first of 2 consecutive visits with plasma HIV-1 RNA greater than or equal to 40 copies/milliliter (mL), if the participant previously demonstrated 2 consecutive plasma HIV-1 RNA levels below 40 copies/mL; Study Day 1, if the subject never achieved 2 consecutive plasma HIV-1 RNA levels below 40 copies/mL; the day of the final measurement, if the final measurement was the first one documenting an increase in plasma HIV-1 RNA level to greater than or equal to 40 copies/mL.
Time Frame: Baseline to Week 96
Population: Intent to treat (ITT) population, defined as all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 105 | 101
Percentage of Participants | 79.1 | 77.8

7. Secondary Outcome: Number of Participants Who Developed Resistance to Each Drug in the Study Regimen, as Defined by the International AIDS Society-USA (IAS-USA) Panel.
Description: Resistance to study drugs was defined as described by the International AIDS Society-USA (IAS-USA) Panel. All participants had an HIV-1 drug resistance genotype (lopinavir/ritonavir, tenofovir, or emtricitabine) obtained at the Screening Visit. Beginning at Week 8, if participant's plasma HIV-1 RNA was greater than or equal to 40 copies/milliliter (mL) and was below 40 copies/mL at the previous visit, additional procedures were undertaken to determine if resistance to study drug occurred.
Time Frame: Baseline to Week 96
Population: The population for each group was the number of participants who met the criteria for resistance testing, that is, participants whose HIV-RNA increased from <40 copies/ml to >=40 copies/mL at a later visit and who underwent additional genotyping for resistance to one of the study drugs the participant was receiving.
Measure: Number; unit: Participants
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 5 | 8
Participants
  Lopinavir resistance | 0 | 0
  Emtricitabine resistance | 1 | 0
  Tenofovir resistance | 0 | 0
  Raltegravir resistance | NA — Participants in this treatment group did not receive raltegravir; as a result, the potential for developing resistance to raltegravir is not applicable. | 3

8. Secondary Outcome: Number of Participants Who Developed Resistance, Defined Conservatively, to Lopinavir
Description: Beginning at Week 8, if participant's plasma HIV-1 RNA was greater than/equal to 40 copies/milliliter (mL) and was below 40 copies/mL at the previous visit, additional procedures were undertaken to determine if resistance occurred. Evidence of lopinavir resistance was more conservatively defined as the presence of 1 or more of these mutations: protease I47V or A, G48V, I50V, V82A or F or T or S, I84V, L90M; or presence of at least 3 or more of these mutations: protease L10F or I or R or V, K20M or R, L24I, V32I, L33F, M36I, M46I or L, F53L, any change to I54, A71V or T, and G73S.
Time Frame: Baseline to Week 96
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 5 | 8
Participants | 0 | 1

9. Secondary Outcome: Change From Baseline on Physical Component Score of the Medical Outcomes Study HIV Health Survey
Description: The Survey is a brief, comprehensive health status measure used in studies of people with HIV/AIDS. Participants rate their health and mental/emotional condition, how much their health limits physical activities (eating, dressing, bathing, climbing stairs, walking one block, etc.) and social activities (for example, visiting with friends or relatives), and other questions that measure quality of life. The physical component summarizes answers to questions about physical status. Possible scores range from 0 to 100. A higher score indicates better health, and increases indicate improvement.
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 75 | 67
Scores on a scale | -1.0 (1.34) | -1.1 (1.51)

10. Secondary Outcome: Change From Baseline on Mental Component of Medical Outcomes Study HIV Health Survey
Description: The Survey is a brief, comprehensive health status measure used in studies of people with HIV/AIDS. Participants rate their health and mental/emotional condition, how much their health limits physical activities (eating, dressing, bathing, climbing stairs, walking one block, etc.) and social activities (visiting with friends or relatives, etc.), and other questions that measure quality of life. The mental component summarizes answers to questions about emotional and mental wellbeing. Possible scores range from 0 to 100. Higher scores indicates better health, and increases indicate improvement.
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 75 | 67
Scores on a scale | 1.3 (1.44) | 1.3 (1.62)

11. Secondary Outcome: Score on Effectiveness Scale of Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: The Effectiveness Scale of the TSQM evaluates the participant's satisfaction or dissatisfaction (1=extremely dissatisfied to 7=extremely satisfied) with the ability of the medication to prevent or treat the condition, the way the medication relieves symptoms, the amount of time it takes for the medication to start working, and other questions. Scores are converted to a range of 0 to 100. A higher score indicates greater satisfaction.
Time Frame: Week 96
Population: Participants who had values at Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 84 | 80
Scores on a scale | 75.5 (23.29) | 76.0 (27.47)

12. Secondary Outcome: Score on Side Effects Scale of Treatment Satisfaction Questionnaire for Medication
Description: The Side Effects scale of the TSQM asks if the participant experiences side effects (yes/no), and if so, how bothersome the side effects are, to what extent they interfere with physical health and ability to function (for example, strength and energy levels), to what extent they interfere with mental function (for example, ability to think clearly, stay awake, etc.), and to what extent the side effects affect the participants overall satisfaction with the medication. Scores are converted to a range of 0 to 100. Higher scores indicate less interference and/or less dissatisfaction.
Time Frame: Week 96
Population: Participants who had values at Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 85 | 80
Scores on a scale | 84.6 (17.56) | 86.2 (19.15)

13. Secondary Outcome: Score on Global Satisfaction Scale of Treatment Satisfaction Questionnaire for Medication
Description: The Global Satisfaction scale of the TSQM evaluates the participants rating of whether the good things about the medication outweigh the bad things (1=not at all certain to 5=extremely certain) and how satisfied or dissatisfied the participant is with the medication (1=extremely dissatisfied to 7=extremely satisfied). Scores are converted to a range of 0 to 100. Higher scores indicate greater satisfaction.
Time Frame: Week 96
Population: Participants who had values at Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 85 | 80
Scores on a scale | 82.5 (15.49) | 85.5 (15.62)

14. Secondary Outcome: Mean Change From Baseline in Hemoglobin (Grams/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 88 | 82
grams/liter | 5.4 (13.26) | 5.1 (13.05)

15. Secondary Outcome: Mean Change From Baseline in Hematocrit (Fraction)
Description: Hematocrit fraction is the percentage (%) by volume of packed red blood cells (RBCs) in the participant's blood. It was measured using standard clinical laboratory analysis of participants' blood samples.
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: % by volume of packed RBCs in blood
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 88 | 82
% by volume of packed RBCs in blood | 0.038 (0.0379) | 0.036 (0.0386)

16. Secondary Outcome: Mean Change From Baseline in Red Blood Cell Count (x 10^12/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: number of cells x 10^12/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 88 | 82
number of cells x 10^12/liter | 0.12 (0.450) | 0.16 (0.471)

17. Secondary Outcome: Mean Change From Baseline in Platelet Count (x 10^9/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: number of cells x 10^9/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 88 | 82
number of cells x 10^9/liter | 46.8 (69.18) | 34.2 (68.94)

18. Secondary Outcome: Mean Change From Baseline in White Blood Cell Count (x 10^9/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: number of cells x 10^9/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 88 | 82
number of cells x 10^9/liter | 0.90 (1.717) | 1.20 (1.670)

19. Secondary Outcome: Mean Change From Baseline in Neutrophils (x 10^9/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: number of cells x 10^9/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 88 | 82
number of cells x 10^9/liter | 0.509 (1.2256) | 0.705 (1.2836)

20. Secondary Outcome: Mean Change From Baseline in Lymphocytes (x 10^9/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: number of cells x 10^9/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 88 | 82
number of cells x 10^9/liter | 0.332 (0.6901) | 0.368 (0.8068)

21. Secondary Outcome: Mean Change From Baseline in Monocytes (x 10^9/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: number of cells x 10^9/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 88 | 82
number of cells x 10^9/liter | 0.065 (0.1435) | 0.112 (0.1436)

22. Secondary Outcome: Mean Change From Baseline in Eosinophils (x 10^9/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: number of cells x 10^9/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 88 | 82
number of cells x 10^9/liter | -0.012 (0.0817) | 0.015 (0.1063)

23. Secondary Outcome: Mean Change From Baseline in Basophils (x 10^9/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: number of cells x 10^9/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 88 | 82
number of cells x 10^9/liter | 0.005 (0.0233) | 0.003 (0.0222)

24. Secondary Outcome: Mean Change From Baseline in Alanine Aminotransferase (Units/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
units/liter | -6.1 (41.45) | -13.4 (39.96)

25. Secondary Outcome: Mean Change From Baseline in Aspartate Aminotransferase (Units/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
units/liter | -0.8 (64.29) | -9.6 (37.86)

26. Secondary Outcome: Mean Change From Baseline in Alkaline Phosphatase (Units/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
units/liter | 14.5 (20.26) | 1.7 (24.53)

27. Secondary Outcome: Mean Change From Baseline in Creatine Phosphokinase (Units/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
units/liter | 398.9 (3381.10) | 157.2 (1081.24)

28. Secondary Outcome: Mean Change From Baseline in Total Bilirubin (Micromoles/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
micromoles/liter | 0.9 (4.17) | 1.9 (6.16)

29. Secondary Outcome: Mean Change From Baseline in Creatinine (Micromoles/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
micromoles/liter | 5.7 (12.66) | 1.6 (11.54)

30. Secondary Outcome: Mean Change From Baseline in Blood Urea Nitrogen (Micromoles/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
micromoles/liter | 0.00 (1.390) | 0.37 (1.658)

31. Secondary Outcome: Mean Change From Baseline in Uric Acid (Micromoles/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
micromoles/liter | -29.0 (65.25) | -6.1 (66.29)

32. Secondary Outcome: Mean Change From Baseline in Inorganic Phosphate (Micromoles/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
micromoles/liter | -0.046 (0.1645) | -0.028 (0.2391)

33. Secondary Outcome: Mean Change From Baseline in Calcium (Micromoles/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
micromoles/liter | -0.040 (0.1071) | -0.016 (0.1468)

34. Secondary Outcome: Mean Change From Baseline in Sodium (Micromoles/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
micromoles/liter | 0.1 (2.04) | 0.7 (2.49)

35. Secondary Outcome: Mean Change From Baseline in Potassium (Micromoles/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
micromoles/liter | 0.13 (0.386) | 0.03 (0.386)

36. Secondary Outcome: Mean Change From Baseline in Chloride (Micromoles/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
micromoles/liter | -0.4 (2.51) | 0.2 (3.65)

37. Secondary Outcome: Mean Change From Baseline in Bicarbonate (Micromoles/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
micromoles/liter | -0.5 (2.79) | -0.8 (3.28)

38. Secondary Outcome: Mean Change From Baseline in Albumin (Grams/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
grams/liter | 1.4 (3.48) | 1.3 (3.66)

39. Secondary Outcome: Mean Change From Baseline in Total Protein (Grams/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
grams/liter | -6.3 (6.07) | -7.2 (6.80)

40. Secondary Outcome: Mean Change From Baseline in Cholesterol (Micromoles/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
micromoles/liter | 0.808 (1.0327) | 1.113 (1.1699)

41. Secondary Outcome: Mean Change From Baseline in High Density Lipoprotein Cholesterol (HDL) (Micromoles/Liter)
Description: Included in measures of metabolic toxicity
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
micromoles/liter | 0.257 (0.3060) | 0.346 (0.3162)

42. Secondary Outcome: Mean Change From Baseline in Low Density Lipoprotein (LDL) (Micromoles/Liter)
Description: Included in measures of metabolic toxicity
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
micromoles/liter | 0.535 (0.8583) | 0.715 (0.9831)

43. Secondary Outcome: Mean Change From Baseline in Low Density Lipoprotein (LDL): High Density Lipoprotein (HDL) Ratio (Ratio)
Time Frame: Baseline to Week 96
Population: Participants who had values for both measures (LDL and HDL) at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
ratio | -0.056 (0.7798) | -0.040 (0.9119)

44. Secondary Outcome: Mean Change From Baseline in Triglycerides (Micromoles/Liter)
Description: Included in measures of metabolic toxicity
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
micromoles/liter | 0.846 (1.5874) | 1.103 (1.6805)

45. Secondary Outcome: Mean Change From Baseline in Calculated Creatinine Clearance (Milliliters/Second)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: milliliters/second
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
milliliters/second | -0.122 (0.3047) | -0.024 (0.3020)

46. Secondary Outcome: Mean Change From Baseline in Fasting Glucose (Millimoles/Liter)
Description: Included in measures of metabolic toxicity
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: millimoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 80
millimoles/liter | -0.011 (0.7501) | 0.109 (1.1172)

47. Secondary Outcome: Mean Change From Baseline in Lactate Dehydrogenase (Units/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 89 | 81
units/liter | -21.157 (69.2920) | -28.926 (41.4161)

48. Secondary Outcome: Mean Change From Baseline in Lipase (Units/Liter)
Description: Included in measures of metabolic toxicity
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
units/liter | 4.674 (54.3370) | -1.898 (24.5716)

49. Secondary Outcome: Mean Change From Baseline in Magnesium (Millimoles/Liter)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: millimoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
millimoles/liter | 0.019 (0.0748) | -0.009 (0.0763)

50. Secondary Outcome: Mean Change From Baseline in Adiponectin (Micrograms/Milliliter)
Description: Included in measures of metabolic toxicity
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 89 | 78
micrograms/milliliter | 2.112 (7.3600) | 2.064 (4.9970)

51. Secondary Outcome: Mean Change From Baseline in Interleukin-6 (Nanograms/Liter)
Description: Included in measures of metabolic toxicity
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: nanograms/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 89 | 77
nanograms/liter | -1.584 (9.4362) | -53.286 (422.1502)

52. Secondary Outcome: Mean Change From Baseline in Lactate (Millimoles/Liter)
Description: Included in measures of metabolic toxicity
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: millimoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 86 | 74
millimoles/liter | 0.281 (0.6456) | 0.444 (1.2115)

53. Secondary Outcome: Mean Change From Baseline in Soluble Tumor Necrosis Factor Receptor-1 (Picograms/Milliliter)
Description: Included in measures of metabolic toxicity
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: picograms/milliliter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 88 | 77
picograms/milliliter | -138.602 (362.1327) | -166.403 (482.2808)

54. Secondary Outcome: Mean Change From Baseline in Soluble Tumor Necrosis Factor Receptor-2 (Picograms/Milliliter)
Description: Included in measures of metabolic toxicity
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: picograms/milliliter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 88 | 77
picograms/milliliter | -1257.9 (1354.75) | -1594.7 (1682.78)

55. Secondary Outcome: Mean Change From Baseline in Leptin (Nanograms/Milliliter)
Description: Included in measures of metabolic toxicity
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 88 | 78
nanograms/milliliter | 3.623 (7.3797) | 2.927 (6.4420)

56. Secondary Outcome: Mean Change From Baseline in Insulin (Picomoles/Liter)
Description: Included in measures of metabolic toxicity
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: picomoles/liter
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 91 | 81
picomoles/liter | -6.724 (49.2087) | 4.441 (72.8859)

57. Secondary Outcome: Mean Change From Baseline in Urine Specific Gravity
Description: Urine specific gravity is a laboratory test that measures the concentration of all chemical particles in the urine. The measurement produces a ratio of the urine density to water density.
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: ratio of urine density to water density
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 83 | 77
ratio of urine density to water density | 0.0042 (0.00742) | 0.0052 (0.00746)

58. Secondary Outcome: Mean Change From Baseline in Urine pH
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 83 | 77
pH | 0.00 (0.672) | 0.03 (0.819)

59. Secondary Outcome: Mean Change From Baseline in Sitting Systolic Blood Pressure (mm Hg)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
mm Hg | -0.7 (16.45) | -2.4 (15.20)

60. Secondary Outcome: Mean Change From Baseline in Sitting Diastolic Blood Pressure (mm Hg)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
mm Hg | -2.4 (9.96) | -1.8 (10.56)

61. Secondary Outcome: Mean Change From Baseline in Sitting Heart Rate (Beats Per Minute)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 88 | 79
beats per minute | -4.6 (13.30) | -6.3 (13.72)

62. Secondary Outcome: Mean Change From Baseline in Weight (kg)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 82
kg | 1.83 (7.106) | 3.77 (6.781)

63. Secondary Outcome: Mean Change From Baseline in Temperature (°F)
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: °F
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 77
°F | -0.152 (0.8069) | -0.183 (0.8768)

64. Secondary Outcome: Mean Change From Baseline in Chest Measurement (cm)
Description: Chest circumference is included in the measures of somatic toxicity, which is characterized by loss of fat in the face, arms, and legs, and increase in fat in the base of the back of the neck and in the abdomen. Participant's chest circumference was measured at 5 cm above the xiphoid process using non-stretchable measuring tape with half centimeter marks.
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 were included in the analysis.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 91 | 84
cm | 1.13 (6.010) | 4.06 (18.903)

65. Secondary Outcome: Mean Change From Baseline in Waist Measurement (cm)
Description: Waist circumference is included in the measures of somatic toxicity, which is characterized by loss of fat in the face, arms, and legs, and increase in fat in the base of the back of the neck and in the abdomen. Circumference of participant's waist was measured at the level of the navel using non-stretchable measuring tape with half centimeter marks.
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 92 | 84
cm | 1.88 (8.489) | 4.93 (20.344)

66. Secondary Outcome: Mean Change From Baseline in Mid-Arm Measurement (cm)
Description: Arm circumference is included in the measures of somatic toxicity, which is characterized by loss of fat in the face, arms, and legs, and increase in fat in the base of the back of the neck and in the abdomen. Particpant's arm circumference was measured halfway between the acromial process on the shoulder and the tip of the elbow (olecranon process) using non-stretchable measuring tape with half centimeter marks.
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 92 | 84
cm | 1.76 (19.688) | 4.71 (20.844)

67. Secondary Outcome: Mean Change From Baseline in Hips Measurement (cm)
Description: Hip circumference is included in the measures of somatic toxicity, which is characterized by loss of fat in the face, arms, and legs, and increase in fat in the base of the back of the neck and in the abdomen. Participant was measured at widest width of the hip using non-stretchable measuring tape with half centimeter marks.
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 92 | 84
cm | 2.45 (7.565) | 4.70 (18.784)

68. Secondary Outcome: Mean Change From Baseline in Mid-Thigh Measurement (cm)
Description: Mid-thigh circumference is included in the measures of somatic toxicity, which is characterized by loss of fat in the face, arms, and legs, and increase in fat in the base of the back of the neck and in the abdomen. Particpant's thigh circumference was measured halfway between the inguinal crease and the midpoint of the upper border of the patella using non-stretchable measuring tape with half centimeter marks.
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 90 | 84
cm | 2.09 (21.148) | 5.13 (25.969)

69. Secondary Outcome: Mean Change From Baseline in Dual Energy X-ray Absorptiometry (DEXA) Scan of Upper Extremity Fat (Grams)
Description: The dual energy X-ray absorptiometry (DEXA) scan is included in the measures of somatic toxicity, which is characterized by loss of fat in the face, arms, and legs, and increase in fat in the base of the back of the neck and in the abdomen.
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 78
grams | 7.28 (31.953) | 21.53 (52.911)

70. Secondary Outcome: Mean Change From Baseline in Dual Energy X-ray Absorptiometry (DEXA) Scan of Upper Extremity Lean Mass (Grams)
Description: as for outcome 69
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 78
grams | -1.49 (7.725) | -1.25 (10.693)

71. Secondary Outcome: Mean Change From Baseline in Dual Energy X-ray Absorptiometry (DEXA) Scan of Upper Extremity Total Mass (Grams)
Description: as for outcome 69
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 78
grams | -0.33 (9.013) | 1.52 (12.911)

72. Secondary Outcome: Mean Change From Baseline in Dual Energy X-ray Absorptiometry (DEXA) Scan of Lower Extremity Fat (Grams)
Description: The dual energy X-ray absorptiometry (DEXA) is included in the measures of somatic toxicity, which is characterized by loss of fat in the face, arms, and legs, and increase in fat in the base of the back of the neck and in the abdomen.
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 78
grams | 15.32 (31.250) | 28.82 (49.855)

73. Secondary Outcome: Mean Change From Baseline in DEXA Scan of Lower Extremity Lean Mass (Grams)
Description: as for outcome 69
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 78
grams | 1.97 (6.220) | 2.27 (8.080)

74. Secondary Outcome: Mean Change From Baseline in Dual Energy X-ray Absorptiometry (DEXA) Scan of Lower Extremity Total Mass (Grams)
Description: as for outcome 69
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 78
grams | 4.32 (9.797) | 6.96 (11.466)

75. Secondary Outcome: Mean Change From Baseline in Dual Energy X-ray Absorptiometry (DEXA) Scan of Trunk Fat (Grams)
Description: as for outcome 69
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 78
grams | 13.75 (40.009) | 27.01 (65.086)

76. Secondary Outcome: Mean Change From Baseline in Dual Energy X-ray Absorptiometry (DEXA) Scan of Trunk Lean Mass (Grams)
Description: as for outcome 69
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 78
grams | 1.67 (5.988) | 2.56 (7.248)

77. Secondary Outcome: Mean Change From Baseline in Dual Energy X-ray Absorptiometry (DEXA) Scan of Trunk Mass (Grams)
Description: as for outcome 69
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 78
grams | 3.48 (9.352) | 6.34 (10.122)

78. Secondary Outcome: Mean Change From Baseline in Dual Energy X-ray Absorptiometry (DEXA) Scan of Total Body Fat (Grams)
Description: as for outcome 69
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 78
grams | 12.71 (33.543) | 25.31 (53.892)

79. Secondary Outcome: Mean Change From Baseline in Dual Energy X-ray Absorptiometry (DEXA) Scan of Total Body Lean Mass (Grams)
Description: as for outcome 69
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 78
grams | 1.08 (5.224) | 1.56 (6.005)

80. Secondary Outcome: Mean Change From Baseline in Dual Energy X-ray Absorptiometry (DEXA) Scan of Total Body Mass (Grams)
Description: as for outcome 69
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 78
grams | 2.9 (8.52) | 5.4 (9.42)

81. Secondary Outcome: Mean Change From Baseline in Dual Energy X-ray Absorptiometry (DEXA) Scan of Bone Mineral Content (Grams)
Description: The dual energy X-ray absorptiometry (DEXA) scan of bone mineral content was used to evaluate potential bone effects of treatment.
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 78
grams | -3.69 (5.224) | 0.52 (5.861)

82. Secondary Outcome: Mean Change From Baseline in Dual Energy X-ray Absorptiometry (DEXA) Scan of Bone Mineral Density (Grams/cm^2)
Description: as for outcome 81
Time Frame: Baseline to Week 96
Population: Participants who had values at Baseline and Week 96 are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams/cm^2
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Number analyzed (Participants) | 82 | 78
grams/cm^2 | -2.48 (3.797) | 0.68 (4.614)

ADVERSE EVENTS:
Time Frame: Week 96
Description: Treatment-emergent adverse events were defined as those occurring after study drug initiation and within 30 days after the last dose of study drug.
Arm/Group | LPV/r + FTC/TDF | LPV/r + RAL
Serious Adverse Events (participants affected / at risk) | 14/105 | 12/101
Other Adverse Events (participants affected / at risk) | 96/105 | 94/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LPV/r + FTC/TDF (N=105) | LPV/r + RAL (N=101)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Anogenital warts (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 2 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Drug abuse (Psychiatric disorders) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Infected sebaceous cyst (Infections and infestations) | 1 | 0
Lymphogranuloma venereum (Infections and infestations) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1
Proctocolitis (Gastrointestinal disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Scrotal infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 2
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Typhoid fever (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LPV/r + FTC/TDF (N=105) | LPV/r + RAL (N=101)
Abdominal pain (Gastrointestinal disorders) | 10 | 4
Anogenital warts (Infections and infestations) | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 8
Asthenia (General disorders) | 8 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 6
Bronchitis (Infections and infestations) | 11 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Depression (Psychiatric disorders) | 11 | 10
Diarrhoea (Gastrointestinal disorders) | 64 | 62
Dizziness (Nervous system disorders) | 7 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 6
Fatigue (General disorders) | 7 | 4
Flatulence (Gastrointestinal disorders) | 9 | 11
Folliculitis (Infections and infestations) | 1 | 7
Gastroenteritis (Infections and infestations) | 6 | 5
Headache (Nervous system disorders) | 18 | 13
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 | 15
Hypertension (Vascular disorders) | 6 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | 16
Influenza (Infections and infestations) | 4 | 8
Insomnia (Psychiatric disorders) | 10 | 9
Nasopharyngitis (Infections and infestations) | 15 | 11
Nausea (Gastrointestinal disorders) | 20 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Pharyngitis (Infections and infestations) | 4 | 6
Pyrexia (General disorders) | 9 | 6
Rash (Skin and subcutaneous tissue disorders) | 4 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Sinusitis (Infections and infestations) | 8 | 6
Syphilis (Infections and infestations) | 5 | 6
Upper respiratory tract infection (Infections and infestations) | 10 | 14
Urinary tract infection (Infections and infestations) | 8 | 3
Vertigo (Ear and labyrinth disorders) | 3 | 6
Vomiting (Gastrointestinal disorders) | 13 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.